CLINICAL TRIAL: NCT05329727
Title: The Comparative Effectiveness Study Between ARNI and ACE Inhibitor/ARB Medication in Patient With Heart Failure With Reduced Ejection Fraction Using the Nationwide Population Based Real World Registry of Korean Heart Failure
Brief Title: The Comparative Effectiveness Between ARNI and ACE Inhibitor/ARB Medication in Patient With HFrEF
Acronym: PARADE-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Byung-Su Yoo, Professor, Wonju Severance Christian Hospital
Other Study IDs: CR321358
Record Dates: First submitted 2022-04-07; First posted 2022-04-15 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure; Mortality
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Angiotensin receptor neprilysin inhibitor (ARNI) — The group with ARNI was defined as patients with HFrEF took ARNI more than 3 months
  Other Names: ARNI
Drug: Renin-Angiotensin System Inhibitor (RAS inhibitor) — The group with RAS inhibitor was defined as patients with HFrEF took RAS inhibitor more than 3 months
  Other Names: RAS inhibitor

SUMMARY:
This study aimed to evaluate the effectiveness, safety, and cost-effectiveness of ARNI and ACEi/ARBs in real-world practice. This study could find out what the unmet medical needs are in real world practice. Furthermore, this study will be helpful to establish the healthcare policy reimbursement policy or clinical practice guideline for HF regarding HF medications to reduce the burden of HF in Korea.

DETAILED DESCRIPTION:
Despite developments and improvements in treatment strategies, heart failure (HF) remains a significant socioeconomic burden and leads to individual health problems due to its high mortality and readmission rates. The latest 2016 European Society of Cardiology (ESC) guideline recommends pharmacological treatment indicated in patients with symptomatic HF with reduced ejection fraction. As the Class I level, the ESC guideline recommends 'ACEI, ARB, ARNI, BB, MRA, Diuretics'. Guideline-directed medication therapy (GDMT) significantly improved the survival of HF, particularly heart failure with reduced ejection fraction (HFrEF). However, various registry studies demonstrated that HFrEF patients are frequently undertreated. The gap exists between the ideal guideline and the current practice of HF treatment. According to the observational nationwide study using the Korean National Health Insurance Claims database, still, 28.6% of elderly heart failure patients did not receive evidence-based treatment. To reduce the various burdens of HF at the patient and society level, the right understanding of the disease and a nationwide systematic approach are needed.

Recently, more data have emerged to support an expanded role for ARNIs in patients with HFrEF. These data include their use as a de novo therapy in some patients naive to ACEIs or ARB therapies, evidence for rapid improvement in patient-reported outcome measures, and the demonstration of a reverse-remodeling effect of ARNIs in chronic HFrEF, independent of background therapy with ACEIs/ARBs. However, the use of ARNI is still under expectation. Clinical trials showed a fabulous result with the use of ARNI in HFrEF patients, however, real-world data is still lacking. In Korea, the use of ARNI is increasing, however, the exact use of ARNI is unknown, and only limited data reported the prescription pattern and outcomes of ARNI in HFrEF patients.

Korea has an obligatory public health insurance system, the term of the Korean National Health Insurance Service (NHIS) with which more than 97% of people are affiliated. All claim data is electronically recorded and can be investigated for research purposes with the approval of the Research Ethics Committee. The use of medications, dosage, cost, and the effect on HF outcomes are assessable using the Korean NHIS database. Previous studies about HF using the NHIS database have several limitations. They were conducted in small research groups, and the operational definition of each study was different, and no studies were conducted after sufficient discussions with HF expert opinions from the Korean Society of Heart Failure.

This study aimed to evaluate the effectiveness, safety, and cost-effectiveness of ARNI and ACEi/ARBs in real-world practice. This study could find out what the unmet medical needs are in real-world practice. Furthermore, this study will be helpful to establish the healthcare policy reimbursement policy or clinical practice guidelines for HF regarding HF medications to reduce the burden of HF in Korea.

This is a non-interventional retrospective cohort study. This study will collect primary data and secondary use data. The data will originate from the NHIS database. Clinical characteristics (age, sex, BMI, WC, lipid profile, LFT, physical activity) will be investigated. The treatment patterns are to be summarized using the proportion of patients with good guideline adherence. Finally, it will compare the clinical outcomes (hospitalization rate, cardiovascular and all-cause mortality) and medical costs of patients groups who were treated with ARNI and without ARNI.

This study will collect primary data and secondary use data in patients with HF between 2017 and 2021. Data sources might include socioeconomic status, abstracts of primary clinical records, electronic medical records, prescription drug files, laboratory reports, and questionnaires for health behaviors. Concomitant or prior medications entered into the database will be coded using the NHIS Reference List. Medical history/current medical conditions will be coded using ICD-10 codes.

The Kaplan-Meier will be used for the survival curve to analyze the primary endpoints (all-cause mortality, CV mortality, or first/recurrent any hospitalization ) and the related results. Normally distributed continuous data are reported as mean ± standard deviation, while non-parametric data are reported as median with interquartile range in brackets. Categorical data are reported as numbers with percentages in brackets. Comparisons between continuous variables were made using independent t-tests, while chi-square tests were made for comparisons between categorical variables, with posthoc correction for tests including more than two groups. Propensity score matching (maximum 1:5) will be performed for those who had used ARNI and those who had not (ACEi/ARBs). The propensity score analysis balances covariates between study groups of observational data using a propensity score, which is the conditional probability of assignment to a particular group given observed covariates only. The investigators will derive the propensity score model from a multiple logistic regression that included age, sex, and underlying comorbidities. A stratified Cox proportional hazards regression model for matched data will be used to evaluate the relation between the treatments and study outcomes (mortality and/or first/recurrent any hospitalization).

ELIGIBILITY:
Inclusion Criteria:

* HF patients were defined as those with "heart failure" according to the disease code in the main code and the sub-code in the claims data.

HF patients who were assigned the following KCD-6 disease codes were considered as: "hypertensive heart disease with (congestive) HF" (I11.0), "hypertensive heart and renal disease with (congestive) HF" (I13.0), "hypertensive heart and renal disease with both (congestive) HF and renal failure" (I13.2), and "HF" (I50) including "congestive HF" (I50.0), "LV failure" (I50.1), and "HF and unspecified" (I50.9).

* HFrEF patients were defined with the following KCD-6 disease codes: "Congestive heart failure with systolic dysfunction"(I5004), "Left ventricular failure"(I501), "Ischaemic cardiomyopathy"(I22.5), "Dilated cardiomyopathy" (I420).

Hospitalized heart failure is defined as the HF disease code and admission.

Exclusion Criteria:

* Less than 18 years old
* In case where investigators determine it's inappropriate to be included in the study as per investigators' clinical judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HF patients with new use of ARNI will be 1:1 propensity score matched with HF patients without ARNI use. Cohort entry was the day of the first filled prescription of ARNI. Study participants were patients aged 18 years or older with HF, which is, with an inpatient or outpatient HF diagnosis recorded during the year prior to drug initiation.
Sampling Method: Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence rate (%) of composite endpoint including all-cause mortality or hospital readmission | 12 months
  all cause mortality: death due to any cause.
  Hospital readmission: any readmission
The medical cost (won) of medical care | 12 months
  The total medical cost of hospitalization due to HF and visitation to the outpatients clinic due to HF

CONTACTS AND LOCATIONS:
Overall Officials: Byung Su Yoo, MD,PhD, Principal Investigator — Yonsei Wonju Christian Hospital
Locations (1):
- Yonsei University Wonju College of Medicine, Wŏnju, Gangwondo, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsao CW, Lyass A, Enserro D, Larson MG, Ho JE, Kizer JR, Gottdiener JS, Psaty BM, Vasan RS. Temporal Trends in the Incidence of and Mortality Associated With Heart Failure With Preserved and Reduced Ejection Fraction. JACC Heart Fail. 2018 Aug;6(8):678-685. doi: 10.1016/j.jchf.2018.03.006. Epub 2018 Jul 11. PMID 30007560
- [Background] Cho DH, Yoo BS. Current Prevalence, Incidence, and Outcomes of Heart Failure with Preserved Ejection Fraction. Heart Fail Clin. 2021 Jul;17(3):315-326. doi: 10.1016/j.hfc.2021.03.002. PMID 34051964
- [Background] Chang PP, Wruck LM, Shahar E, Rossi JS, Loehr LR, Russell SD, Agarwal SK, Konety SH, Rodriguez CJ, Rosamond WD. Trends in Hospitalizations and Survival of Acute Decompensated Heart Failure in Four US Communities (2005-2014): ARIC Study Community Surveillance. Circulation. 2018 Jul 3;138(1):12-24. doi: 10.1161/CIRCULATIONAHA.117.027551. Epub 2018 Mar 8. PMID 29519849
- [Background] Conrad N, Judge A, Tran J, Mohseni H, Hedgecott D, Crespillo AP, Allison M, Hemingway H, Cleland JG, McMurray JJV, Rahimi K. Temporal trends and patterns in heart failure incidence: a population-based study of 4 million individuals. Lancet. 2018 Feb 10;391(10120):572-580. doi: 10.1016/S0140-6736(17)32520-5. Epub 2017 Nov 21. PMID 29174292
- [Background] Lee JH, Lim NK, Cho MC, Park HY. Epidemiology of Heart Failure in Korea: Present and Future. Korean Circ J. 2016 Sep;46(5):658-664. doi: 10.4070/kcj.2016.46.5.658. Epub 2016 Sep 28. PMID 27721857
- [Background] Choi EK. Cardiovascular Research Using the Korean National Health Information Database. Korean Circ J. 2020 Sep;50(9):754-772. doi: 10.4070/kcj.2020.0171. Epub 2020 May 20. PMID 32725984
- [Derived] Cho DH, Choi J, Youn JC, Kim MN, Lee CJ, Son JW, Yoo BS. Angiotensin receptor-neprilysin inhibitor adherence and outcomes in heart failure with reduced ejection fraction. ESC Heart Fail. 2025 Feb;12(1):603-612. doi: 10.1002/ehf2.15117. Epub 2024 Oct 17. PMID 39420468